CLINICAL TRIAL: NCT02610257
Title: The Role of Somatosensory Dysfunction as the Underlying Mechanism of Upper Limbs Motor Blocks in People With Parkinson's Disease With and Without Freezing of Gait
Brief Title: Somatosensory Dysfunction as the Underlying Mechanism of Upper Limbs Motor Blocks in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Alice Nieuwboer, Full professor Faculty of Kinesiology and Rehabilitation Sciences, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: S58674
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease; Somatosensory Disorders
Keywords: Parkinson's disease; Freezing of gait; Motor blocks; Somatosensory; Proprioception; Muscle vibration; Handwriting
MeSH Terms: conditions — Parkinson Disease; Somatosensory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vibration Relevant (Active Comparator): Vibration applied on the muscle belly after 'motor block' onset
  Interventions: Device: Mechanical stimulus (vibration) applied on the forearm
- Neutral Vibration Relevant (Active Comparator): Vibration applied on a bony mark after 'motor block' onset
  Interventions: Device: Mechanical stimulus (vibration) applied on the forearm
- Neutral Vibration Non-Relevant (Active Comparator): Vibration applied on a bony mark before 'motor block' onset
  Interventions: Device: Mechanical stimulus (vibration) applied on the forearm
- Vibration Non-Relevant (Active Comparator): Vibration applied on the muscle belly after 'motor block' onset
  Interventions: Device: Mechanical stimulus (vibration) applied on the forearm
- No Vibration (No Intervention)

INTERVENTIONS:
Device: Mechanical stimulus (vibration) applied on the forearm — Local vibration will be applied using a custom-made vibratory system (named Vibrators) consisted of small vibratory devices (constructed using DC micro motors (Faulhaber® - Switzerland) bearing an eccentric load, enclosure on a PVC involucre). Vibrators measure 4.5cm x 2cm x 2cm and weight 27-31g each. Vibrators were custom-made especially for this study and therefore do not have a trade name.
  Vibrators will be positioned either on the extensor carpi radialis brevis (ECRB) muscle belly or on the olecranon region. Devices will be kept in place using regular elbow elastic supports.
  Arms: Neutral Vibration Non-Relevant; Neutral Vibration Relevant; Vibration Non-Relevant; Vibration Relevant

SUMMARY:
Motor blocks during gait and upper limb movements (FOULs) are a disabling and common motor impairment in mild to severe stages of Parkinson's disease (PD). However, the main mechanism underlying these phenomena is still an open debate. Apart from the motor correlates, cognitive-attentional impairment and somatosensory deficits (especially in the proprioceptive system) may underlie these motor blocks. The current study aims to unravel whether the proprioceptive system is involved by manipulating task-relevant or non-relevant proprioceptive stimuli.

Hence, the main aims of this study are:

(i) to assess the somatosensory function in people with PD that experience freezing of gait FOG and (ii) to investigate the effects of manipulating both proprioception and attentional resources on FOUL severity.

Forty-five people will be assigned to three age-matched groups (N=15 each): healthy elderly, PD patients that experience FOG (FOG+) and PD patients that do not experience FOG. Cutaneous sensory function and kinesthetic ability will be assessed by means of standardized user-friendly methods and precise repositioning measures using the VICON motion analysis. Additionally, participants will perform a newly developed task that can successfully elicit FOULs (a handwriting freezing-provoking task) on a custom tablet (Heremans et al 2015). The task will be performed without and with the use of muscle vibration (a well-known method to stimulate the proprioceptive system). The investigators will manipulate both the timing of vibration (relevant - after FOUL onset; or non-relevant: before FOUL onset) and the region of stimulation (neutral: on a bone-mark where there is little if any proprioceptive stimulation; and on a non-neutral spot: on the forearm muscles). It is believed that FOG+ will present with worse somatosensory function than those who do not experience motor blocks (especially in the proprioceptive system). Additionally, the Investigators expect a reduction in FOUL severity (e.g. FOUL duration) when vibration is applied in a task-relevant way, independently of the region stimulated. In contrast, it is also expected that when vibration is applied in a non-relevant way and it may act as a distractor, FOUL duration will increase. This study will thus be able to distinguish between the contribution of attentional and proprioceptive resources to the mechanism of motor blocks in PD.

ELIGIBILITY:
Inclusion Criteria:

* PD patients (N=30):
* Diagnosis of PD based on the UK PD brain bank criteria
* Hoehn & Yahr stage II-III (ON-medication)

Exclusion Criteria:

* Cognitive dysfunction Score on the Mini Mental State Examination (MMSE) < 23/30
* Medication change in the past 1 month
* Other neurological disorders
* Vestibular disorder
* Uncontrolled diabetes
* Cutaneous diseases
* Left-handedness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in upper limb motor blocks duration | 30 min
Joint Position Sense | 15 min
  Participants will be comfortably seated, while both forearms rest on a table with hands facing down. Then, the right arm should slowly and actively be moved to a certain target angle indicated by the test leader. This target angle should be memorized while holding their arm at this position for 4s, after which participants slowly return their arm to the starting position. After 3s, participants will be asked to actively reproduce the previous target position with the same limb. All trials will be conducted while participants maintain their eyes closed and with their elbow off the table surface. The limb position will be recorded by using 7 MX-T20 optoelectronic cameras (Vicon, Oxford Metrics, UK). For this 3D movement analysis, each participant will be instrumented with 10 spherical reflective markers positioned on participants' right shoulder, arm, elbow, forearm and hand.
Perceptual Threshold of Touch | 15 min
  For this test a dual channel nerve stimulator (TENS) will be used (CEFAR PRIMO PRO - CEFAR Medical AB®). Participants will be seated in a standardized and comfortable way, allowing them to observe the entire procedure. Two individual electrodes (3cm of diameter) will be placed on bulb of the index finger (anode) and on the tenar region of the same limb (cathode). A constant current of 40Hz with single square pulses with 80μs of duration will be used. The current amplitude will be increased in steps of 0.5mA at every 2 seconds. The participant will be instructed to say "now" when they feel a slight tingling sensation. Three trials will be used for both hands. The Perceptual Threshold of Touch will be considered as the average of the three trials. It is expected that subjects will feel a slight itching and painless sensation. To avoid any discomfort, the test will be interrupted whenever an involuntary movement is seen, since the Motor Threshold always precedes the Pain Threshold.

SECONDARY OUTCOMES:
Writing amplitude assessed by a tablet | 30 min
  The paradigm consists of performing a task on a 16.5cm length tablet (Fujitsu Componentes Europe®) .The device is powered by a regular laptop. To maximize participants' comfort the tablet screen is squared. The task consists of a 'freezing-provoking task'. This 'freezing-provoking' task has already been tested in people with PD in a current writing study at the Neuromotor Research Group . This task has been shown to be highly successful to elicit motor blocks in the upper limbs in PD patients (data submitted for publication). Each trial will last 30 seconds and as much trials as needed will be provided before the data collection to ensure participants have learned the task.
Somatosensory Function | 30 min
  Assessed by the Erasmus Notthingham Sensory Assessment (EmNSA)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, Professor, Principal Investigator — KU Leuven
Locations (1):
- CatholicULeuven, Leuven, Belgium

REFERENCES:
- See also: Related Info — http://gbiomed.kuleuven.be/english/research/50000743/nrrg1/nr.htm